CLINICAL TRIAL: NCT00430300
Title: A Phase II, Randomized, Double Blind, Placebo Controlled, Parallel Group Study To Evaluate the Efficacy And Safety of UK-432,097 Dry Powder For Inhalation In Adults With Moderate To Severe Chronic Obstructive Pulmonary Disease.
Brief Title: Safety And Efficacy Of UK-432,097 In Chronic Obstructive Pulmonary Disease.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3971013
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Results first posted 2013-07-08 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Dry Powder for Inhalation; Chronic Obstructive Pulmonary Disease; Lung Function testing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 150mcg, 450mcg or 1350mcg (Experimental): Active treatment given BID via a double pin monodose capsule inhaler device
  Interventions: Drug: UK-432,097
- Placebo (Placebo Comparator): Placebo treatment given BID via a single pin monodose inhaler device
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UK-432,097 — Formulated as a dry powder, supplied as capsules and administered using an atomizer device. Given as either 150mcg, 450mcg or 1350mcg BID.
  Arms: 150mcg, 450mcg or 1350mcg
Drug: Placebo — Capsules containing 100% lactose administered BID using an atomizer device
  Arms: Placebo

SUMMARY:
Safety and efficacy (measured by spirometry) of UK-432,097 administration will be tested in patients with chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis, for at least 6 months, of moderate to severe COPD (GOLD) and who meet the criteria for Stage II-III disease
* Patients must have a smoking history of at least 10 pack-years
* Patients must have stable disease for at least 1 month prior to screening.

Exclusion Criteria:

* More than 2 exacerbations of COPD in the preceding year
* History of a lower respiratory tract infection or significant disease instability during the month proceding screening or during the time between screen and randomization.
* History or presence of respiratory failure, cor pulmonale or right ventricular failure

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- Australia (4):
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Glebe, New South Wales
  - Pfizer Investigational Site, Daw Park, South Australia
  - Pfizer Investigational Site, Nedlands, Western Australia
- Canada (5):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Trois-Rivières, Quebec
- Netherlands (3):
  - Pfizer Investigational Site, Almelo
  - Pfizer Investigational Site, Eindhoven
  - Pfizer Investigational Site, Zuthpen
- Poland (4):
  - Pfizer Investigational Site, Bydgoszcz, Poland
  - Pfizer Investigational Site, Gdansk, Poland
  - Pfizer Investigational Site, Warsaw, Poland
  - Pfizer Investigational Site, Lodz
- United Kingdom (6):
  - Pfizer Investigational Site, Chertsey, Surrey
  - Pfizer Investigational Site, Leicester
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Newcastle upon Tyne
  - Pfizer Investigational Site, Southampton

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3971013&StudyName=Safety%20And%20Efficacy%20Of%20UK-432%2C097%20In%20Chronic%20Obstructive%20Pulmonary%20Disease.

RESULTS

PARTICIPANT FLOW:
Groups:
- UK-432,097 150 Mcg: UK-432,097 150 microgram (mcg) capsule and 2 matching placebo capsules twice daily up to Week 6, administered by inhalation using the single pin mono-dose capsule inhaler device. Additionally, participants received ipratropium bromide metered dose inhaler (MDI) 2 actuations (20 mcg/actuation) 4 times daily as a maintenance therapy up to Week 8 and salbutamol MDI 1 to 2 actuations (100 mcg/actuation) as rescue therapy whenever required.
- UK-432,097 450 Mcg: UK-432,097 450 mcg capsule and 2 matching placebo capsules twice daily up to Week 6, administered by inhalation using the single pin mono-dose capsule inhaler device. Additionally, participants received ipratropium bromide MDI 2 actuations (20 mcg/actuation) 4 times daily as a maintenance therapy up to Week 8 and salbutamol MDI 1 to 2 actuations (100 mcg/actuation) as rescue therapy whenever required.
- UK-432,097 1350 Mcg: UK-432,097 1350 mcg (3 * 450 mcg capsules) twice daily up to Week 6, administered by inhalation using the single pin mono-dose capsule inhaler device. Additionally, participants received ipratropium bromide MDI 2 actuations (20 mcg/actuation) 4 times daily as a maintenance therapy up to Week 8 and salbutamol MDI 1 to 2 actuations (100 mcg/actuation) as rescue therapy whenever required.
- Placebo: Placebo matching to UK-432,097 capsules twice daily up to Week 6, administered by inhalation using the single pin mono-dose capsule inhaler device. Additionally, participants received ipratropium bromide MDI 2 actuations (20 mcg/actuation) 4 times daily as a maintenance therapy up to Week 8 and salbutamol MDI 1 to 2 actuations (100 mcg/actuation) as rescue therapy whenever required.
Period: Overall Study
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Started | 17 | 18 | 35 | 17
Completed | 15 | 16 | 29 | 15
Not Completed | 2 | 2 | 6 | 2
Not completed — Adverse Event | 0 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 5 | 0
Not completed — Laboratory abnormality | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- UK-432,097 150 Mcg: UK-432,097 150 mcg capsule and 2 matching placebo capsules twice daily up to Week 6, administered by inhalation using the single pin mono-dose capsule inhaler device. Additionally, participants received ipratropium bromide MDI 2 actuations (20 mcg/actuation) 4 times daily as a maintenance therapy up to Week 8 and salbutamol MDI 1 to 2 actuations (100 mcg/actuation) as rescue therapy whenever required.
- Total: Total of all reporting groups
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo | Total
Number analyzed (Participants) | 17 | 18 | 35 | 17 | 87
Age, Customized [Number; unit: participants]
  45 to 64 Years | 8 | 7 | 12 | 9 | 36
  Greater Than or Equal to (>=) 65 Years | 9 | 11 | 23 | 8 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 9 | 6 | 25
  Male | 12 | 13 | 26 | 11 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 6
Description: FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Trough FEV1 was obtained from spirometry, performed before study treatment administration.
Time Frame: Pre-dose at Baseline, Week 6
Population: Full analysis set (FAS): all randomized participants, who received at least 2 weeks of dosing and had at least 1 valid FEV1 measurement during treatment. Missing data were imputed using Last Observation Carried Forward (LOCF). Here 'n' signifies participants who were evaluable for this measure at specified time-point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 16 | 17 | 32 | 16
liter
  Baseline (n= 16, 17, 32, 16) | 1.40 (0.45) | 1.48 (0.57) | 1.41 (0.39) | 1.33 (0.48)
  Change at Week 6 (n= 14, 17, 29, 15) | -0.01 (0.21) | -0.05 (0.18) | -0.05 (0.18) | -0.05 (0.16)
Statistical Analysis 1: Comparison: UK-432,097 150 Mcg vs Placebo; The Bayesian normal dynamic linear model (NDLM) was used for analysis. 95% credible intervals of the effect size and the posterior distribution were calculated. Posterior distribution was used to calculate a probability (presented as p value) that the dose gives a difference of 0.075 liter from placebo; Test type: Superiority or Other; p = 0.0284, Bayesian NDLM model; NDLM estimate difference = -0.0087, 95% CI 2-sided [-0.0943 to 0.0774]
Statistical Analysis 2: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0056, Bayesian NDLM model; NDLM estimate difference = -0.0389, 95% CI 2-sided [-0.1299 to 0.0471]
Statistical Analysis 3: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0009, Bayesian NDLM model; NDLM estimate difference = -0.0510, 95% CI 2-sided [-0.1298 to 0.0290]

2. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 2, 4 and 8
Description: as for outcome 1
Time Frame: Pre-dose at Baseline, Week 2, 4, 8
Population: FAS: all randomized participants, who received at least 2 weeks of dosing and had at least 1 valid FEV1 measurement during treatment. Here 'n' signifies participants who were evaluable for this measure at specified time-point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 16 | 17 | 32 | 16
liter
  Change at Week 2 (n= 16, 17, 32, 16) | -0.01 (0.10) | -0.10 (0.11) | 0.01 (0.13) | 0.01 (0.18)
  Change at Week 4 (n= 15, 17, 30, 16) | -0.08 (0.19) | -0.06 (0.15) | -0.02 (0.17) | -0.01 (0.12)
  Change at Week 8 (n= 14, 16, 27, 16) | 0.03 (0.23) | -0.07 (0.18) | 0.04 (0.23) | -0.05 (0.17)
Statistical Analysis 1: Comparison: UK-432,097 150 Mcg vs Placebo; Change at Week 2: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.5849, Mixed Models Analysis; Adjusted Mean Difference = -0.01, 95% CI 1-sided [lower limit -0.09], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9737, Mixed Models Analysis; Adjusted Mean Difference = -0.09, 95% CI 1-sided [lower limit -0.17], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3870, Mixed Models Analysis; Adjusted Mean Difference = 0.01, 95% CI 1-sided [lower limit -0.06], Standard Error of Mean 0.04
Statistical Analysis 4: Comparison: UK-432,097 150 Mcg vs Placebo; Change at Week 4: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.8612, Mixed Models Analysis; Adjusted Mean Difference = -0.06, 95% CI 1-sided [lower limit -0.15], Standard Error of Mean 0.06
Statistical Analysis 5: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.7499, Mixed Models Analysis; Adjusted Mean Difference = -0.04, 95% CI 1-sided [lower limit -0.13], Standard Error of Mean 0.05
Statistical Analysis 6: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.5134, Mixed Models Analysis; Adjusted Mean Difference = -0.00, 95% CI 1-sided [lower limit -0.08], Standard Error of Mean 0.05
Statistical Analysis 7: Comparison: UK-432,097 150 Mcg vs Placebo; Change at Week 8: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.1244, Mixed Models Analysis; Adjusted Mean Difference = 0.08, 95% CI 1-sided [lower limit -0.04], Standard Error of Mean 0.07
Statistical Analysis 8: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.5300, Mixed Models Analysis; Adjusted Mean Difference = -0.01, 95% CI 1-sided [lower limit -0.12], Standard Error of Mean 0.07
Statistical Analysis 9: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.0550, Mixed Models Analysis; Adjusted Mean Difference = 0.10, 95% CI 1-sided [lower limit -0.00], Standard Error of Mean 0.06

3. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 6 Seconds (FEV6) at Week 2, 4, 6 and 8
Description: FEV6 is the maximal volume of air exhaled in the first 6 seconds of a forced expiration from a position of full inspiration. Trough FEV6 was obtained from spirometry, performed before study treatment administration.
Time Frame: Pre-dose at Baseline, Week 2, 4, 6, 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 16 | 17 | 32 | 16
liter
  Baseline (n= 16, 17, 32, 16) | 2.66 (0.73) | 2.80 (0.81) | 2.75 (0.69) | 2.54 (0.73)
  Change at Week 2 (n= 16, 17, 32, 16) | -0.02 (0.22) | -0.08 (0.18) | -0.01 (0.20) | 0.03 (0.19)
  Change at Week 4 (n= 15, 17, 30, 16) | -0.12 (0.24) | 0.03 (0.19) | -0.05 (0.23) | -0.01 (0.13)
  Change at Week 6 (n= 14, 17, 29, 15) | -0.00 (0.25) | 0.01 (0.30) | -0.06 (0.22) | -0.05 (0.18)
  Change at Week 8 (n= 14, 16, 27, 16) | 0.10 (0.34) | -0.05 (0.31) | 0.04 (0.30) | -0.09 (0.26)
Statistical Analysis 1: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7444, Mixed Models Analysis; Adjusted Mean Difference = -0.05, 95% CI 1-sided [lower limit -0.16], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9134, Mixed Models Analysis; Adjusted Mean Difference = -0.10, 95% CI 1-sided [lower limit -0.21], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6841, Mixed Models Analysis; Adjusted Mean Difference = -0.03, 95% CI 1-sided [lower limit -0.13], Standard Error of Mean 0.06
Statistical Analysis 4: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.9283, Mixed Models Analysis; Adjusted Mean Difference = -0.11, 95% CI 1-sided [lower limit -0.23], Standard Error of Mean 0.07
Statistical Analysis 5: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.2991, Mixed Models Analysis; Adjusted Mean Difference = 0.04, 95% CI 1-sided [lower limit -0.08], Standard Error of Mean 0.07
Statistical Analysis 6: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.7403, Mixed Models Analysis; Adjusted Mean Difference = -0.04, 95% CI 1-sided [lower limit -0.15], Standard Error of Mean 0.06
Statistical Analysis 7: Comparison: UK-432,097 150 Mcg vs Placebo; Change at Week 6: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.3499, Mixed Models Analysis; Adjusted Mean Difference = 0.03, 95% CI 1-sided [lower limit -0.11], Standard Error of Mean 0.09
Statistical Analysis 8: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.2734, Mixed Models Analysis; Adjusted Mean Difference = 0.05, 95% CI 1-sided [lower limit -0.09], Standard Error of Mean 0.08
Statistical Analysis 9: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.5806, Mixed Models Analysis; Adjusted Mean Difference = -0.02, 95% CI 1-sided [lower limit -0.14], Standard Error of Mean 0.07
Statistical Analysis 10: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.0540, Mixed Models Analysis; Adjusted Mean Difference = 0.18, 95% CI 1-sided [lower limit -0.00], Standard Error of Mean 0.11
Statistical Analysis 11: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.2616, Mixed Models Analysis; Adjusted Mean Difference = 0.07, 95% CI 1-sided [lower limit -0.11], Standard Error of Mean 0.10
Statistical Analysis 12: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.0724, Mixed Models Analysis; Adjusted Mean Difference = 0.14, 95% CI 1-sided [lower limit -0.02], Standard Error of Mean 0.09

4. Secondary Outcome: Change From Baseline in Trough Forced Vital Capacity (FVC) at Week 2, 4, 6 and 8
Description: FVC is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Trough FVC was obtained from spirometry, performed before study treatment administration.
Time Frame: Pre-dose at Baseline, Week 2, 4, 6, 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 16 | 17 | 32 | 16
liter
  Baseline (n= 16, 17, 32, 16) | 3.11 (0.85) | 3.43 (1.16) | 3.24 (0.91) | 3.01 (0.94)
  Change at Week 2 (n= 16, 17, 32, 16) | -0.07 (0.30) | -0.09 (0.30) | -0.04 (0.25) | 0.09 (0.31)
  Change at Week 4 (n= 15, 17, 30, 16) | -0.14 (0.34) | 0.14 (0.21) | -0.02 (0.32) | 0.05 (0.21)
  Change at Week 6 (n= 14, 17, 29, 15) | 0.01 (0.32) | 0.01 (0.33) | -0.01 (0.31) | 0.02 (0.17)
  Change at Week 8 (n= 14, 16, 27, 16) | 0.14 (0.46) | 0.02 (0.40) | 0.07 (0.33) | -0.05 (0.28)
Statistical Analysis 1: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9362, Mixed Models Analysis; Adjusted Mean Difference = -0.15, 95% CI 1-sided [lower limit -0.32], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9469, Mixed Models Analysis; Adjusted Mean Difference = -0.16, 95% CI 1-sided [lower limit -0.33], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9153, Mixed Models Analysis; Adjusted Mean Difference = -0.12, 95% CI 1-sided [lower limit -0.27], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.9686, Mixed Models Analysis; Adjusted Mean Difference = -0.19, 95% CI 1-sided [lower limit -0.36], Standard Error of Mean 0.10
Statistical Analysis 5: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.1548, Mixed Models Analysis; Adjusted Mean Difference = 0.10, 95% CI 1-sided [lower limit -0.06], Standard Error of Mean 0.10
Statistical Analysis 6: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.7973, Mixed Models Analysis; Adjusted Mean Difference = -0.07, 95% CI 1-sided [lower limit -0.22], Standard Error of Mean 0.09
Statistical Analysis 7: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.6348, Mixed Models Analysis; Adjusted Mean Difference = -0.04, 95% CI 1-sided [lower limit -0.22], Standard Error of Mean 0.11
Statistical Analysis 8: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.5742, Mixed Models Analysis; Adjusted Mean Difference = -0.02, 95% CI 1-sided [lower limit -0.19], Standard Error of Mean 0.10
Statistical Analysis 9: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.6719, Mixed Models Analysis; Adjusted Mean Difference = -0.04, 95% CI 1-sided [lower limit -0.19], Standard Error of Mean 0.09
Statistical Analysis 10: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.0881, Mixed Models Analysis; Adjusted Mean Difference = 0.18, 95% CI 1-sided [lower limit -0.04], Standard Error of Mean 0.13
Statistical Analysis 11: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.2772, Mixed Models Analysis; Adjusted Mean Difference = 0.07, 95% CI 1-sided [lower limit -0.13], Standard Error of Mean 0.12
Statistical Analysis 12: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.1363, Mixed Models Analysis; Adjusted Mean Difference = 0.12, 95% CI 1-sided [lower limit -0.06], Standard Error of Mean 0.11

5. Secondary Outcome: Change From Baseline in Trough Inspiratory Capacity (IC) at Week 2, 4, 6 and 8
Description: IC is the maximum volume of air that can be inhaled into the lungs from the normal resting position after breathing out normally. Trough IC was obtained from spirometry, performed before study treatment administration.
Time Frame: Pre-dose at Baseline, Week 2, 4, 6, 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 16 | 17 | 32 | 16
liter
  Baseline (n= 16, 17, 32, 16) | 2.44 (0.63) | 2.81 (0.78) | 2.53 (0.59) | 2.41 (0.82)
  Change at Week 2 (n= 16, 17, 32, 16) | 0.03 (0.27) | -0.06 (0.38) | -0.03 (0.30) | -0.10 (0.24)
  Change at Week 4 (n= 15, 17, 30, 16) | -0.05 (0.18) | -0.03 (0.38) | -0.15 (0.28) | -0.06 (0.25)
  Change at Week 6 (n= 14, 17, 29, 15) | -0.03 (0.23) | -0.08 (0.40) | -0.14 (0.28) | -0.09 (0.32)
  Change at Week 8 (n= 14, 16, 27, 16) | 0.07 (0.22) | 0.01 (0.44) | -0.10 (0.33) | -0.05 (0.26)
Statistical Analysis 1: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0938, Mixed Models Analysis; Adjusted Mean Difference = 0.14, 95% CI 1-sided [lower limit -0.03], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2149, Mixed Models Analysis; Adjusted Mean Difference = 0.08, 95% CI 1-sided [lower limit -0.09], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1682, Mixed Models Analysis; Adjusted Mean Difference = 0.09, 95% CI 1-sided [lower limit -0.06], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.4492, Mixed Models Analysis; Adjusted Mean Difference = 0.01, 95% CI 1-sided [lower limit -0.16], Standard Error of Mean 0.10
Statistical Analysis 5: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.2539, Mixed Models Analysis; Adjusted Mean Difference = 0.07, 95% CI 1-sided [lower limit -0.10], Standard Error of Mean 0.10
Statistical Analysis 6: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.8168, Mixed Models Analysis; Adjusted Mean Difference = -0.08, 95% CI 1-sided [lower limit -0.22], Standard Error of Mean 0.09
Statistical Analysis 7: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.3248, Mixed Models Analysis; Adjusted Mean Difference = 0.05, 95% CI 1-sided [lower limit -0.13], Standard Error of Mean 0.11
Statistical Analysis 8: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.3148, Mixed Models Analysis; Adjusted Mean Difference = 0.05, 95% CI 1-sided [lower limit -0.13], Standard Error of Mean 0.11
Statistical Analysis 9: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.6563, Mixed Models Analysis; Adjusted Mean Difference = -0.04, 95% CI 1-sided [lower limit -0.20], Standard Error of Mean 0.09
Statistical Analysis 10: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.1735, Mixed Models Analysis; Adjusted Mean Difference = 0.12, 95% CI 1-sided [lower limit -0.09], Standard Error of Mean 0.12
Statistical Analysis 11: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.1237, Mixed Models Analysis; Adjusted Mean Difference = 0.14, 95% CI 1-sided [lower limit -0.06], Standard Error of Mean 0.12
Statistical Analysis 12: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.6113, Mixed Models Analysis; Adjusted Mean Difference = -0.03, 95% CI 1-sided [lower limit -0.21], Standard Error of Mean 0.11

6. Secondary Outcome: Change From Baseline in Post-Study Drug FEV1 at Week 2, 4, and 6
Description: FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Post-study drug FEV1 was obtained from spirometry, performed 15-30 minutes after study treatment administration.
Time Frame: 15 to 30 minutes post-dose at Baseline, Week 2, 4, 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 16 | 17 | 32 | 16
liter
  Baseline (n= 16, 17, 32, 16) | 1.40 (0.45) | 1.48 (0.57) | 1.41 (0.39) | 1.33 (0.48)
  Change at Week 2 (n= 16, 16, 30, 16) | 0.02 (0.11) | -0.10 (0.16) | -0.02 (0.11) | 0.03 (0.20)
  Change at Week 4 (n= 14, 16, 29, 16) | -0.07 (0.15) | -0.04 (0.10) | -0.02 (0.15) | -0.01 (0.15)
  Change at Week 6 (n= 13, 16, 27, 15) | -0.06 (0.23) | -0.04 (0.18) | -0.04 (0.15) | -0.03 (0.20)
Statistical Analysis 1: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5549, Mixed Models Analysis; Adjusted Mean Difference = -0.01, 95% CI 1-sided [lower limit -0.09], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9880, Mixed Models Analysis; Adjusted Mean Difference = -0.11, 95% CI 1-sided [lower limit -0.20], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8572, Mixed Models Analysis; Adjusted Mean Difference = -0.05, 95% CI 1-sided [lower limit -0.12], Standard Error of Mean 0.04
Statistical Analysis 4: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.8402, Mixed Models Analysis; Adjusted Mean Difference = -0.05, 95% CI 1-sided [lower limit -0.14], Standard Error of Mean 0.05
Statistical Analysis 5: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.6562, Mixed Models Analysis; Adjusted Mean Difference = -0.02, 95% CI 1-sided [lower limit -0.10], Standard Error of Mean 0.05
Statistical Analysis 6: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.5632, Mixed Models Analysis; Adjusted Mean Difference = -0.01, 95% CI 1-sided [lower limit -0.08], Standard Error of Mean 0.04
Statistical Analysis 7: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.6370, Mixed Models Analysis; Adjusted Mean Difference = -0.02, 95% CI 1-sided [lower limit -0.13], Standard Error of Mean 0.07
Statistical Analysis 8: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.4686, Mixed Models Analysis; Adjusted Mean Difference = 0.01, 95% CI 1-sided [lower limit -0.10], Standard Error of Mean 0.06
Statistical Analysis 9: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.6164, Mixed Models Analysis; Adjusted Mean Difference = -0.02, 95% CI 1-sided [lower limit -0.11], Standard Error of Mean 0.06

7. Secondary Outcome: Change From Baseline in Post-Study Drug FEV6 at Week 2, 4, and 6
Description: FEV6 is the maximal volume of air exhaled in the first 6 seconds of a forced expiration from a position of full inspiration. Post-study drug FEV6 was obtained from spirometry, performed 15-30 minutes after study treatment administration.
Time Frame: 15 to 30 minutes post-dose at Baseline, Week 2, 4, 6
Population: Data for this pre-specified outcome was not analyzed, as the study was terminated due to futility based on results of interim analysis.
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Post-Study Drug FVC at Week 2, 4, and 6
Description: FVC is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Post-study drug FVC was obtained from spirometry, performed 15-30 minutes after study treatment administration.
Time Frame: 15 to 30 minutes post-dose at Baseline, Week 2, 4, 6
Population: as for outcome 7
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Post-Study Drug IC at Week 2, 4, and 6
Description: IC is the maximum amount of air that can be inhaled into the lungs from the normal resting position after breathing out normally. Post-study drug IC was obtained from spirometry, performed 15-30 minutes after study treatment administration.
Time Frame: 15 to 30 minutes post-dose at Baseline, Week 2, 4, 6
Population: as for outcome 7
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Change From Baseline in Post-Bronchodilator FEV1 at Week 6
Description: FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Post-bronchodilator FEV1 was obtained from spirometry, performed 15-30 minutes after bronchodilator (salbutamol) administration.
Time Frame: 15 to 30 minutes post-bronchodilator administration at Baseline, Week 6
Population: FAS: all randomized participants, who received at least 2 weeks of dosing and had at least 1 valid FEV1 measurement during treatment. Here 'N'(number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 13 | 16 | 27 | 14
liter
  Baseline | 0.32 (0.20) | 0.29 (0.19) | 0.26 (0.18) | 0.24 (0.15)
  Change at Week 6 | 0.06 (0.14) | 0.03 (0.19) | -0.02 (0.19) | -0.06 (0.14)

11. Secondary Outcome: Change From Baseline in Post-Bronchodilator FEV6 at Week 6
Description: FEV6 is the maximal volume of air exhaled in the first 6 seconds of a forced expiration from a position of full inspiration. Post-bronchodilator FEV6 was obtained from spirometry, performed 15-30 minutes after bronchodilator (salbutamol) administration.
Time Frame: 15 to 30 minutes post-bronchodilator administration at Baseline, Week 6
Population: as for outcome 7
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in Post-Bronchodilator FVC at Week 6
Description: FVC is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Post-bronchodilator FVC was obtained from spirometry, performed 15-30 minutes after bronchodilator (salbutamol) administration.
Time Frame: 15 to 30 minutes post-bronchodilator administration at Baseline, Week 6
Population: as for outcome 7
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Change From Baseline in Post-Bronchodilator IC at Week 6
Description: IC is the maximum volume of air that can be inhaled into the lungs from the normal resting position after breathing out normally. Post-bronchodilator IC was obtained from spirometry, performed 15-30 minutes after bronchodilator (salbutamol) administration.
Time Frame: 15 to 30 minutes post-bronchodilator administration at Baseline, Week 6
Population: as for outcome 7
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Change From Baseline in Dyspnea (Baseline Dyspnea Index/Transition Dyspnea Index [BDI/TDI]) at Week 2, 4, and 6
Description: BDI: 24-item questionnaire to assess baseline dyspnea in 3 domains, functional impairment; magnitude of task; magnitude of effort. Each item rated on 5-point scale: 0 (very severe), 4 (no impairment). BDI total score range: 0 to 12, lower score=more severe dyspnea. TDI: 24-item questionnaire to measure changes in dyspnea severity from baseline in same 3 domains, as in BDI. Each item rated on 7-point scale: -3 (major deterioration) to 3 (major improvement). TDI total score range: -9 to 9, lower score=more deterioration. BDI/TDI total scores were obtained by adding scores for each of 3 domains.
Time Frame: Baseline, Week 2, 4, 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 16 | 17 | 32 | 16
units on a scale
  BDI (n= 16, 17, 32, 16) | 7.1 (1.9) | 7.6 (2.1) | 7.2 (2.1) | 7.1 (2.0)
  TDI at Week 2 (n= 16, 17, 32, 16) | -0.2 (1.9) | 0.8 (1.9) | 0.2 (1.1) | 1.3 (2.4)
  TDI at Week 4 (n= 15, 17, 31, 16) | 0.5 (2.8) | 0.2 (1.7) | -0.3 (1.9) | 0.3 (2.2)
  TDI at Week 6 (n= 14, 16, 29, 15) | -0.6 (2.3) | 0.9 (3.1) | 0.1 (2.4) | 1.0 (1.9)
Statistical Analysis 1: Comparison: UK-432,097 150 Mcg vs Placebo; TDI at Week 2: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.9885, Mixed Models Analysis; Adjusted Mean Difference = -1.4, 95% CI 1-sided [lower limit -2.4], Standard Error of Mean 0.6
Statistical Analysis 2: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.8055, Mixed Models Analysis; Adjusted Mean Difference = -0.5, 95% CI 1-sided [lower limit -1.5], Standard Error of Mean 0.6
Statistical Analysis 3: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.9759, Mixed Models Analysis; Adjusted Mean Difference = -1.1, 95% CI 1-sided [lower limit -2.0], Standard Error of Mean 0.5
Statistical Analysis 4: Comparison: UK-432,097 150 Mcg vs Placebo; TDI at Week 4: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.4401, Mixed Models Analysis; Adjusted Mean Difference = 0.1, 95% CI 1-sided [lower limit -1.1], Standard Error of Mean 0.7
Statistical Analysis 5: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority or Other; p = 0.5957, Mixed Models Analysis; Adjusted Mean Difference = -0.2, 95% CI 1-sided [lower limit -1.4], Standard Error of Mean 0.7
Statistical Analysis 6: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 14, analysis 4]; Test type: Superiority or Other; p = 0.8302, Mixed Models Analysis; Adjusted Mean Difference = -0.6, 95% CI 1-sided [lower limit -1.7], Standard Error of Mean 0.6
Statistical Analysis 7: Comparison: UK-432,097 150 Mcg vs Placebo; TDI at Week 6: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.9657, Mixed Models Analysis; Adjusted Mean Difference = -1.6, 95% CI 1-sided [lower limit -3.1], Standard Error of Mean 0.9
Statistical Analysis 8: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.6378, Mixed Models Analysis; Adjusted Mean Difference = -0.3, 95% CI 1-sided [lower limit -1.7], Standard Error of Mean 0.9
Statistical Analysis 9: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.8990, Mixed Models Analysis; Adjusted Mean Difference = -1.0, 95% CI 1-sided [lower limit -2.2], Standard Error of Mean 0.8

15. Secondary Outcome: Change From Baseline in Chronic Obstructive Pulmonary Disease (COPD) Symptom Score at Week 1, 2, 3, 4, 5, 6, 7, and 8
Description: COPD symptom score: participants rated the severity of their COPD symptoms (cough, breathlessness, and sputum production) in daily symptom dairy according to how they felt during the past 24 hours on a 4-point scale ranging from 0 (none) to 3 (severe). A participant's daily score for each symptom was averaged over each week.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8
Population: FAS: all randomized participants, who received at least 2 weeks of dosing and had at least 1 valid FEV1 measurement during treatment. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure and 'n' signifies participants who were evaluable for this measure at specified time-point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 16 | 17 | 31 | 16
units on a scale
  Cough: Baseline (n= 16, 17, 31, 16) | 1.09 (0.50) | 0.77 (0.75) | 1.11 (0.67) | 1.06 (0.61)
  Cough: Change at Week 1 (n= 16, 17, 31, 16) | -0.08 (0.46) | 0.11 (0.48) | 0.07 (0.41) | 0.10 (0.50)
  Cough: Change at Week 2 (n= 16, 15, 31, 16) | -0.10 (0.43) | 0.13 (0.31) | 0.10 (0.53) | -0.01 (0.41)
  Cough: Change at Week 3 (n= 15, 17, 31, 16) | -0.06 (0.51) | 0.15 (0.32) | 0.07 (0.48) | 0.15 (0.41)
  Cough: Change at Week 4 (n= 14, 17, 30, 16) | -0.04 (0.30) | 0.07 (0.38) | -0.03 (0.46) | 0.18 (0.39)
  Cough: Change at Week 5 (n= 15, 17, 30, 16) | -0.13 (0.38) | 0.04 (0.44) | 0.10 (0.73) | 0.00 (0.43)
  Cough: Change at Week 6 (n= 15, 17, 30, 15) | -0.10 (0.36) | 0.04 (0.43) | 0.07 (0.77) | -0.02 (0.40)
  Cough: Change at Week 7 (n= 15, 16, 30, 15) | -0.16 (0.38) | -0.08 (0.57) | 0.00 (0.64) | 0.07 (0.31)
  Cough: Change at Week 8 (n= 15, 16, 28, 15) | -0.15 (0.37) | 0.00 (0.56) | -0.15 (0.60) | 0.07 (0.47)
  Breathlessness: Baseline (n= 16, 17, 31, 16) | 1.31 (0.59) | 1.30 (0.60) | 1.15 (0.75) | 1.27 (0.54)
  Breathlessness: Change at Week 1(n=16, 17, 31, 16) | -0.24 (0.45) | -0.10 (0.31) | -0.05 (0.23) | 0.00 (0.32)
  Breathlessness: Change at Week 2(n=16, 15, 31, 16) | -0.13 (0.48) | -0.11 (0.29) | 0.00 (0.33) | -0.01 (0.38)
  Breathlessness: Change at Week 3(n=15, 17, 31, 16) | -0.12 (0.57) | -0.15 (0.33) | 0.02 (0.33) | 0.13 (0.41)
  Breathlessness: Change at Week 4(n=14, 17, 30, 16) | -0.18 (0.50) | -0.16 (0.50) | -0.07 (0.28) | 0.18 (0.34)
  Breathlessness: Change at Week 5(n=15, 17, 30, 16) | -0.14 (0.47) | -0.22 (0.50) | -0.06 (0.33) | 0.13 (0.40)
  Breathlessness: Change at Week 6(n=15, 17, 30, 15) | -0.12 (0.56) | -0.03 (0.50) | -0.05 (0.34) | 0.12 (0.47)
  Breathlessness: Change at Week 7(n=15, 16, 30, 15) | -0.06 (0.43) | -0.21 (0.48) | 0.01 (0.36) | 0.10 (0.43)
  Breathlessness: Change at Week 8(n=15, 16, 28, 15) | -0.04 (0.49) | -0.13 (0.51) | -0.04 (0.49) | 0.08 (0.45)
  Sputum: Baseline (n= 16, 17, 31, 16) | 1.00 (0.62) | 0.76 (0.79) | 0.95 (0.59) | 0.90 (0.61)
  Sputum: Change at Week 1 (n= 16, 17, 31, 16) | -0.07 (0.26) | 0.10 (0.36) | 0.04 (0.39) | 0.04 (0.41)
  Sputum: Change at Week 2 (n= 16, 15, 31, 16) | -0.05 (0.20) | 0.17 (0.37) | 0.14 (0.54) | 0.05 (0.52)
  Sputum: Change at Week 3 (n= 15, 17, 31, 16) | -0.08 (0.32) | 0.20 (0.37) | 0.15 (0.52) | 0.05 (0.41)
  Sputum: Change at Week 4 (n= 14, 17, 30, 16) | 0.01 (0.21) | 0.15 (0.36) | 0.06 (0.51) | 0.01 (0.47)
  Sputum: Change at Week 5 (n= 15, 17, 30, 16) | 0.06 (0.23) | 0.15 (0.33) | 0.07 (0.48) | -0.04 (0.44)
  Sputum: Change at Week 6 (n= 15, 17, 30, 15) | 0.09 (0.09) | 0.10 (0.46) | 0.10 (0.61) | -0.02 (0.51)
  Sputum: Change at Week 7 (n= 15, 15, 30, 15) | 0.08 (0.23) | -0.02 (0.39) | 0.07 (0.56) | 0.03 (0.51)
  Sputum: Change at Week 8 (n= 15, 15, 28, 15) | 0.07 (0.27) | -0.06 (0.40) | 0.02 (0.47) | -0.03 (0.55)
Statistical Analysis 1: Comparison: UK-432,097 150 Mcg vs Placebo; Cough, Change at Week 1: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.8757, Mixed Models Analysis; Adjusted Mean Difference = -0.17, 95% CI 1-sided [lower limit -0.42], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.6334, Mixed Models Analysis; Adjusted Mean Difference = -0.05, 95% CI 1-sided [lower limit -0.30], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.5448, Mixed Models Analysis; Adjusted Mean Difference = -0.01, 95% CI 1-sided [lower limit -0.23], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: UK-432,097 150 Mcg vs Placebo; Cough, Change at Week 2: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.6986, Mixed Models Analysis; Adjusted Mean Difference = -0.08, 95% CI 1-sided [lower limit -0.34], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 4]; Test type: Superiority or Other; p = 0.3151, Mixed Models Analysis; Adjusted Mean Difference = 0.08, 95% CI 1-sided [lower limit -0.18], Standard Error of Mean 0.16
Statistical Analysis 6: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 4]; Test type: Superiority or Other; p = 0.1802, Mixed Models Analysis; Adjusted Mean Difference = 0.12, 95% CI 1-sided [lower limit -0.10], Standard Error of Mean 0.14
Statistical Analysis 7: Comparison: UK-432,097 150 Mcg vs Placebo; Cough, Change at Week 3: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.9102, Mixed Models Analysis; Adjusted Mean Difference = -0.22, 95% CI 1-sided [lower limit -0.49], Standard Error of Mean 0.16
Statistical Analysis 8: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 7]; Test type: Superiority or Other; p = 0.6391, Mixed Models Analysis; Adjusted Mean Difference = -0.06, 95% CI 1-sided [lower limit -0.32], Standard Error of Mean 0.16
Statistical Analysis 9: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 7]; Test type: Superiority or Other; p = 0.6838, Mixed Models Analysis; Adjusted Mean Difference = -0.07, 95% CI 1-sided [lower limit -0.30], Standard Error of Mean 0.14
Statistical Analysis 10: Comparison: UK-432,097 150 Mcg vs Placebo; Cough, Change at Week 4: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.9648, Mixed Models Analysis; Adjusted Mean Difference = -0.26, 95% CI 1-sided [lower limit -0.49], Standard Error of Mean 0.14
Statistical Analysis 11: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 10]; Test type: Superiority or Other; p = 0.8961, Mixed Models Analysis; Adjusted Mean Difference = -0.17, 95% CI 1-sided [lower limit -0.40], Standard Error of Mean 0.14
Statistical Analysis 12: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 10]; Test type: Superiority or Other; p = 0.9534, Mixed Models Analysis; Adjusted Mean Difference = -0.21, 95% CI 1-sided [lower limit -0.41], Standard Error of Mean 0.12
Statistical Analysis 13: Comparison: UK-432,097 150 Mcg vs Placebo; Cough, Change at Week 5: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.7726, Mixed Models Analysis; Adjusted Mean Difference = -0.14, 95% CI 1-sided [lower limit -0.45], Standard Error of Mean 0.18
Statistical Analysis 14: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.5665, Mixed Models Analysis; Adjusted Mean Difference = -0.03, 95% CI 1-sided [lower limit -0.33], Standard Error of Mean 0.18
Statistical Analysis 15: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.2684, Mixed Models Analysis; Adjusted Mean Difference = 0.10, 95% CI 1-sided [lower limit -0.17], Standard Error of Mean 0.16
Statistical Analysis 16: Comparison: UK-432,097 150 Mcg vs Placebo; Cough, Change at Week 6: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.6485, Mixed Models Analysis; Adjusted Mean Difference = -0.07, 95% CI 1-sided [lower limit -0.39], Standard Error of Mean 0.19
Statistical Analysis 17: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 16]; Test type: Superiority or Other; p = 0.4821, Mixed Models Analysis; Adjusted Mean Difference = 0.01, 95% CI 1-sided [lower limit -0.30], Standard Error of Mean 0.19
Statistical Analysis 18: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 16]; Test type: Superiority or Other; p = 0.2557, Mixed Models Analysis; Adjusted Mean Difference = 0.11, 95% CI 1-sided [lower limit -0.17], Standard Error of Mean 0.16
Statistical Analysis 19: Comparison: UK-432,097 150 Mcg vs Placebo; Cough, Change at Week 7: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.9031, Mixed Models Analysis; Adjusted Mean Difference = -0.23, 95% CI 1-sided [lower limit -0.52], Standard Error of Mean 0.17
Statistical Analysis 20: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 19]; Test type: Superiority or Other; p = 0.8634, Mixed Models Analysis; Adjusted Mean Difference = -0.19, 95% CI 1-sided [lower limit -0.47], Standard Error of Mean 0.17
Statistical Analysis 21: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 19]; Test type: Superiority or Other; p = 0.6375, Mixed Models Analysis; Adjusted Mean Difference = -0.05, 95% CI 1-sided [lower limit -0.30], Standard Error of Mean 0.15
Statistical Analysis 22: Comparison: UK-432,097 150 Mcg vs Placebo; Cough, Change at Week 8: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.8775, Mixed Models Analysis; Adjusted Mean Difference = -0.21, 95% CI 1-sided [lower limit -0.51], Standard Error of Mean 0.18
Statistical Analysis 23: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 22]; Test type: Superiority or Other; p = 0.7191, Mixed Models Analysis; Adjusted Mean Difference = -0.10, 95% CI 1-sided [lower limit -0.40], Standard Error of Mean 0.18
Statistical Analysis 24: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 22]; Test type: Superiority or Other; p = 0.8677, Mixed Models Analysis; Adjusted Mean Difference = -0.18, 95% CI 1-sided [lower limit -0.44], Standard Error of Mean 0.16
Statistical Analysis 25: Comparison: UK-432,097 150 Mcg vs Placebo; Breathlessness, Change at Week 1: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.9838, Mixed Models Analysis; Adjusted Mean Difference = -0.24, 95% CI 1-sided [lower limit -0.42], Standard Error of Mean 0.11
Statistical Analysis 26: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 25]; Test type: Superiority or Other; p = 0.8106, Mixed Models Analysis; Adjusted Mean Difference = -0.10, 95% CI 1-sided [lower limit -0.28], Standard Error of Mean 0.11
Statistical Analysis 27: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 25]; Test type: Superiority or Other; p = 0.7750, Mixed Models Analysis; Adjusted Mean Difference = -0.07, 95% CI 1-sided [lower limit -0.23], Standard Error of Mean 0.10
Statistical Analysis 28: Comparison: UK-432,097 150 Mcg vs Placebo; Breathlessness, Change at Week 2: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.8082, Mixed Models Analysis; Adjusted Mean Difference = -0.11, 95% CI 1-sided [lower limit -0.33], Standard Error of Mean 0.13
Statistical Analysis 29: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 28]; Test type: Superiority or Other; p = 0.7678, Mixed Models Analysis; Adjusted Mean Difference = -0.09, 95% CI 1-sided [lower limit -0.31], Standard Error of Mean 0.13
Statistical Analysis 30: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 28]; Test type: Superiority or Other; p = 0.5373, Mixed Models Analysis; Adjusted Mean Difference = -0.01, 95% CI 1-sided [lower limit -0.20], Standard Error of Mean 0.11
Statistical Analysis 31: Comparison: UK-432,097 150 Mcg vs Placebo; Breathlessness, Change at Week 3: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.9548, Mixed Models Analysis; Adjusted Mean Difference = -0.24, 95% CI 1-sided [lower limit -0.47], Standard Error of Mean 0.14
Statistical Analysis 32: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 31]; Test type: Superiority or Other; p = 0.9743, Mixed Models Analysis; Adjusted Mean Difference = -0.27, 95% CI 1-sided [lower limit -0.49], Standard Error of Mean 0.14
Statistical Analysis 33: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 31]; Test type: Superiority or Other; p = 0.8408, Mixed Models Analysis; Adjusted Mean Difference = -0.12, 95% CI 1-sided [lower limit -0.32], Standard Error of Mean 0.12
Statistical Analysis 34: Comparison: UK-432,097 150 Mcg vs Placebo; Breathlessness, Change at Week 4: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.9887, Mixed Models Analysis; Adjusted Mean Difference = -0.32, 95% CI 1-sided [lower limit -0.55], Standard Error of Mean 0.14
Statistical Analysis 35: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 34]; Test type: Superiority or Other; p = 0.9918, Mixed Models Analysis; Adjusted Mean Difference = -0.33, 95% CI 1-sided [lower limit -0.55], Standard Error of Mean 0.13
Statistical Analysis 36: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 34]; Test type: Superiority or Other; p = 0.9833, Mixed Models Analysis; Adjusted Mean Difference = -0.26, 95% CI 1-sided [lower limit -0.46], Standard Error of Mean 0.12
Statistical Analysis 37: Comparison: UK-432,097 150 Mcg vs Placebo; Breathlessness, Change at Week 5: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.9619, Mixed Models Analysis; Adjusted Mean Difference = -0.26, 95% CI 1-sided [lower limit -0.50], Standard Error of Mean 0.14
Statistical Analysis 38: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 37]; Test type: Superiority or Other; p = 0.9917, Mixed Models Analysis; Adjusted Mean Difference = -0.34, 95% CI 1-sided [lower limit -0.58], Standard Error of Mean 0.14
Statistical Analysis 39: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 37]; Test type: Superiority or Other; p = 0.9376, Mixed Models Analysis; Adjusted Mean Difference = -0.19, 95% CI 1-sided [lower limit -0.40], Standard Error of Mean 0.12
Statistical Analysis 40: Comparison: UK-432,097 150 Mcg vs Placebo; Breathlessness, Change at Week 6: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.9084, Mixed Models Analysis; Adjusted Mean Difference = -0.21, 95% CI 1-sided [lower limit -0.47], Standard Error of Mean 0.16
Statistical Analysis 41: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 40]; Test type: Superiority or Other; p = 0.7906, Mixed Models Analysis; Adjusted Mean Difference = -0.12, 95% CI 1-sided [lower limit -0.38], Standard Error of Mean 0.15
Statistical Analysis 42: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 40]; Test type: Superiority or Other; p = 0.8765, Mixed Models Analysis; Adjusted Mean Difference = -0.16, 95% CI 1-sided [lower limit -0.38], Standard Error of Mean 0.14
Statistical Analysis 43: Comparison: UK-432,097 150 Mcg vs Placebo; Breathlessness, Change at Week 7: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.8469, Mixed Models Analysis; Adjusted Mean Difference = -0.15, 95% CI 1-sided [lower limit -0.38], Standard Error of Mean 0.14
Statistical Analysis 44: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 43]; Test type: Superiority or Other; p = 0.9717, Mixed Models Analysis; Adjusted Mean Difference = -0.27, 95% CI 1-sided [lower limit -0.50], Standard Error of Mean 0.14
Statistical Analysis 45: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 43]; Test type: Superiority or Other; p = 0.7591, Mixed Models Analysis; Adjusted Mean Difference = -0.09, 95% CI 1-sided [lower limit -0.29], Standard Error of Mean 0.12
Statistical Analysis 46: Comparison: UK-432,097 150 Mcg vs Placebo; Breathlessness, Change at Week 8: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.7141, Mixed Models Analysis; Adjusted Mean Difference = -0.10, 95% CI 1-sided [lower limit -0.38], Standard Error of Mean 0.17
Statistical Analysis 47: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 46]; Test type: Superiority or Other; p = 0.8104, Mixed Models Analysis; Adjusted Mean Difference = -0.15, 95% CI 1-sided [lower limit -0.42], Standard Error of Mean 0.17
Statistical Analysis 48: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 46]; Test type: Superiority or Other; p = 0.7664, Mixed Models Analysis; Adjusted Mean Difference = -0.11, 95% CI 1-sided [lower limit -0.35], Standard Error of Mean 0.15
Statistical Analysis 49: Comparison: UK-432,097 150 Mcg vs Placebo; Sputum, Change at Week 1: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.7888, Mixed Models Analysis; Adjusted Mean Difference = -0.10, 95% CI 1-sided [lower limit -0.31], Standard Error of Mean 0.12
Statistical Analysis 50: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 49]; Test type: Superiority or Other; p = 0.3930, Mixed Models Analysis; Adjusted Mean Difference = 0.03, 95% CI 1-sided [lower limit -0.17], Standard Error of Mean 0.12
Statistical Analysis 51: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 49]; Test type: Superiority or Other; p = 0.4785, Mixed Models Analysis; Adjusted Mean Difference = 0.01, 95% CI 1-sided [lower limit -0.17], Standard Error of Mean 0.11
Statistical Analysis 52: Comparison: UK-432,097 150 Mcg vs Placebo; Sputum, Change at Week 2: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.6756, Mixed Models Analysis; Adjusted Mean Difference = -0.07, 95% CI 1-sided [lower limit -0.34], Standard Error of Mean 0.16
Statistical Analysis 53: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 52]; Test type: Superiority or Other; p = 0.2627, Mixed Models Analysis; Adjusted Mean Difference = 0.10, 95% CI 1-sided [lower limit -0.17], Standard Error of Mean 0.16
Statistical Analysis 54: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 52]; Test type: Superiority or Other; p = 0.2281, Mixed Models Analysis; Adjusted Mean Difference = 0.11, 95% CI 1-sided [lower limit -0.13], Standard Error of Mean 0.14
Statistical Analysis 55: Comparison: UK-432,097 150 Mcg vs Placebo; Sputum, Change at Week 3: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.7656, Mixed Models Analysis; Adjusted Mean Difference = -0.12, 95% CI 1-sided [lower limit -0.38], Standard Error of Mean 0.16
Statistical Analysis 56: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 55]; Test type: Superiority or Other; p = 0.2105, Mixed Models Analysis; Adjusted Mean Difference = 0.13, 95% CI 1-sided [lower limit -0.13], Standard Error of Mean 0.16
Statistical Analysis 57: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 55]; Test type: Superiority or Other; p = 0.2221, Mixed Models Analysis; Adjusted Mean Difference = 0.11, 95% CI 1-sided [lower limit -0.12], Standard Error of Mean 0.14
Statistical Analysis 58: Comparison: UK-432,097 150 Mcg vs Placebo; Sputum, Change at Week 4: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.4396, Mixed Models Analysis; Adjusted Mean Difference = 0.02, 95% CI 1-sided [lower limit -0.23], Standard Error of Mean 0.16
Statistical Analysis 59: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 58]; Test type: Superiority or Other; p = 0.2243, Mixed Models Analysis; Adjusted Mean Difference = 0.11, 95% CI 1-sided [lower limit -0.14], Standard Error of Mean 0.15
Statistical Analysis 60: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 58]; Test type: Superiority or Other; p = 0.3597, Mixed Models Analysis; Adjusted Mean Difference = 0.05, 95% CI 1-sided [lower limit -0.17], Standard Error of Mean 0.13
Statistical Analysis 61: Comparison: UK-432,097 150 Mcg vs Placebo; Sputum, Change at Week 5: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.2030, Mixed Models Analysis; Adjusted Mean Difference = 0.12, 95% CI 1-sided [lower limit -0.12], Standard Error of Mean 0.14
Statistical Analysis 62: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 61]; Test type: Superiority or Other; p = 0.1207, Mixed Models Analysis; Adjusted Mean Difference = 0.16, 95% CI 1-sided [lower limit -0.07], Standard Error of Mean 0.14
Statistical Analysis 63: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 61]; Test type: Superiority or Other; p = 0.1836, Mixed Models Analysis; Adjusted Mean Difference = 0.11, 95% CI 1-sided [lower limit -0.09], Standard Error of Mean 0.12
Statistical Analysis 64: Comparison: UK-432,097 150 Mcg vs Placebo; Sputum, Change at Week 6: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.2359, Mixed Models Analysis; Adjusted Mean Difference = 0.12, 95% CI 1-sided [lower limit -0.16], Standard Error of Mean 0.17
Statistical Analysis 65: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 64]; Test type: Superiority or Other; p = 0.2861, Mixed Models Analysis; Adjusted Mean Difference = 0.09, 95% CI 1-sided [lower limit -0.18], Standard Error of Mean 0.17
Statistical Analysis 66: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 64]; Test type: Superiority or Other; p = 0.2151, Mixed Models Analysis; Adjusted Mean Difference = 0.12, 95% CI 1-sided [lower limit -0.13], Standard Error of Mean 0.15
Statistical Analysis 67: Comparison: UK-432,097 150 Mcg vs Placebo; Sputum, Change at Week 7: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.3545, Mixed Models Analysis; Adjusted Mean Difference = 0.06, 95% CI 1-sided [lower limit -0.21], Standard Error of Mean 0.16
Statistical Analysis 68: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 67]; Test type: Superiority or Other; p = 0.7102, Mixed Models Analysis; Adjusted Mean Difference = -0.09, 95% CI 1-sided [lower limit -0.35], Standard Error of Mean 0.16
Statistical Analysis 69: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 67]; Test type: Superiority or Other; p = 0.3883, Mixed Models Analysis; Adjusted Mean Difference = 0.04, 95% CI 1-sided [lower limit -0.19], Standard Error of Mean 0.14
Statistical Analysis 70: Comparison: UK-432,097 150 Mcg vs Placebo; Sputum, Change at Week 8: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.2228, Mixed Models Analysis; Adjusted Mean Difference = 0.12, 95% CI 1-sided [lower limit -0.14], Standard Error of Mean 0.16
Statistical Analysis 71: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 15, analysis 70]; Test type: Superiority or Other; p = 0.6342, Mixed Models Analysis; Adjusted Mean Difference = -0.05, 95% CI 1-sided [lower limit -0.32], Standard Error of Mean 0.16
Statistical Analysis 72: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 15, analysis 70]; Test type: Superiority or Other; p = 0.3141, Mixed Models Analysis; Adjusted Mean Difference = 0.07, 95% CI 1-sided [lower limit -0.16], Standard Error of Mean 0.14

16. Secondary Outcome: Change From Baseline in Rescue Bronchodilator Use at Week 1, 2, 3, 4, 5, 6, 7, and 8
Description: Participants were issued with rescue medication (Salbutamol MDI [100 mcg/actuation]) and were instructed to use 1-2 puffs as required, as a rescue therapy. All rescue medication use was recorded in daily paper dairy by participant. A participant's daily use (puffs/day) was averaged over each week.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: puffs/day
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 14 | 15 | 27 | 15
puffs/day
  Baseline (n= 14, 15, 27, 15) | 2.87 (2.91) | 3.32 (2.99) | 2.97 (2.83) | 3.46 (3.26)
  Change at Week 1 (n= 14, 15, 27, 15) | -0.24 (0.51) | -0.17 (0.53) | -0.19 (0.61) | -0.41 (1.11)
  Change at Week 2 (n= 13, 13, 27, 15) | -0.26 (0.58) | -0.14 (0.67) | -0.08 (0.85) | 0.01 (1.09)
  Change at Week 3 (n= 13, 14, 27, 15) | -0.12 (0.63) | -0.10 (0.79) | 0.03 (0.95) | 0.17 (1.31)
  Change at Week 4 (n= 13, 14, 26, 15) | -0.19 (0.56) | -0.01 (0.99) | -0.08 (0.99) | 0.07 (1.00)
  Change at Week 5 (n= 13, 14, 26, 15) | -0.44 (0.98) | -0.22 (1.39) | 0.21 (1.32) | 0.13 (0.93)
  Change at Week 6 (n= 13, 14, 24, 14) | -0.39 (1.17) | 0.15 (1.16) | 0.26 (1.52) | 0.30 (1.10)
  Change at Week 7 (n= 13, 13, 26, 14) | -0.20 (1.05) | -0.01 (1.81) | 0.38 (1.41) | 0.24 (0.99)
  Change at Week 8 (n= 13, 13, 25, 14) | -0.17 (1.31) | 0.02 (1.51) | 0.30 (1.47) | 0.40 (1.17)
Statistical Analysis 1: Comparison: UK-432,097 150 Mcg vs Placebo; Change at Week 1: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.2700, Mixed Models Analysis; Adjusted Mean Difference = 0.16, 95% CI 1-sided [lower limit -0.28], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.1831, Mixed Models Analysis; Adjusted Mean Difference = 0.24, 95% CI 1-sided [lower limit -0.20], Standard Error of Mean 0.26
Statistical Analysis 3: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.1796, Mixed Models Analysis; Adjusted Mean Difference = 0.21, 95% CI 1-sided [lower limit -0.17], Standard Error of Mean 0.23
Statistical Analysis 4: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8136, Mixed Models Analysis; Adjusted Mean Difference = -0.28, 95% CI 1-sided [lower limit -0.79], Standard Error of Mean 0.31
Statistical Analysis 5: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6877, Mixed Models Analysis; Adjusted Mean Difference = -0.15, 95% CI 1-sided [lower limit -0.66], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6382, Mixed Models Analysis; Adjusted Mean Difference = -0.09, 95% CI 1-sided [lower limit -0.54], Standard Error of Mean 0.27
Statistical Analysis 7: Comparison: UK-432,097 150 Mcg vs Placebo; Change at Week 3: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.7660, Mixed Models Analysis; Adjusted Mean Difference = -0.26, 95% CI 1-sided [lower limit -0.87], Standard Error of Mean 0.36
Statistical Analysis 8: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.7226, Mixed Models Analysis; Adjusted Mean Difference = -0.21, 95% CI 1-sided [lower limit -0.80], Standard Error of Mean 0.35
Statistical Analysis 9: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.6634, Mixed Models Analysis; Adjusted Mean Difference = -0.13, 95% CI 1-sided [lower limit -0.65], Standard Error of Mean 0.31
Statistical Analysis 10: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.7598, Mixed Models Analysis; Adjusted Mean Difference = -0.25, 95% CI 1-sided [lower limit -0.83], Standard Error of Mean 0.35
Statistical Analysis 11: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.5300, Mixed Models Analysis; Adjusted Mean Difference = -0.03, 95% CI 1-sided [lower limit -0.59], Standard Error of Mean 0.34
Statistical Analysis 12: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.7054, Mixed Models Analysis; Adjusted Mean Difference = -0.16, 95% CI 1-sided [lower limit -0.66], Standard Error of Mean 0.30
Statistical Analysis 13: Comparison: UK-432,097 150 Mcg vs Placebo; Change at Week 5: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.8851, Mixed Models Analysis; Adjusted Mean Difference = -0.55, 95% CI 1-sided [lower limit -1.30], Standard Error of Mean 0.45
Statistical Analysis 14: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p = 0.7575, Mixed Models Analysis; Adjusted Mean Difference = -0.31, 95% CI 1-sided [lower limit -1.05], Standard Error of Mean 0.44
Statistical Analysis 15: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p = 0.4325, Mixed Models Analysis; Adjusted Mean Difference = 0.07, 95% CI 1-sided [lower limit -0.58], Standard Error of Mean 0.39
Statistical Analysis 16: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.8934, Mixed Models Analysis; Adjusted Mean Difference = -0.60, 95% CI 1-sided [lower limit -1.41], Standard Error of Mean 0.48
Statistical Analysis 17: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.5283, Mixed Models Analysis; Adjusted Mean Difference = -0.03, 95% CI 1-sided [lower limit -0.82], Standard Error of Mean 0.47
Statistical Analysis 18: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.4900, Mixed Models Analysis; Adjusted Mean Difference = 0.01, 95% CI 1-sided [lower limit -0.68], Standard Error of Mean 0.41
Statistical Analysis 19: Comparison: UK-432,097 150 Mcg vs Placebo; Change at Week 7: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.7465, Mixed Models Analysis; Adjusted Mean Difference = -0.34, 95% CI 1-sided [lower limit -1.20], Standard Error of Mean 0.51
Statistical Analysis 20: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p = 0.5848, Mixed Models Analysis; Adjusted Mean Difference = -0.11, 95% CI 1-sided [lower limit -0.95], Standard Error of Mean 0.51
Statistical Analysis 21: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p = 0.3178, Mixed Models Analysis; Adjusted Mean Difference = 0.21, 95% CI 1-sided [lower limit -0.53], Standard Error of Mean 0.44
Statistical Analysis 22: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.8169, Mixed Models Analysis; Adjusted Mean Difference = -0.47, 95% CI 1-sided [lower limit -1.34], Standard Error of Mean 0.52
Statistical Analysis 23: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.6727, Mixed Models Analysis; Adjusted Mean Difference = -0.23, 95% CI 1-sided [lower limit -1.08], Standard Error of Mean 0.51
Statistical Analysis 24: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.5014, Mixed Models Analysis; Adjusted Mean Difference = -0.00, 95% CI 1-sided [lower limit -0.75], Standard Error of Mean 0.45

17. Secondary Outcome: Change From Baseline in Morning and Evening Peak Expiratory Flow Rate (PEFR) at Week 1, 2, 3, 4, 5, 6, 7, and 8
Description: The PEFR is a participant's maximum speed of expiration, as measured with a peak flow meter. All participants were issued with a hand-held peak flow device and instructed to perform twice daily (morning and evening) prior to taking any medication. A participant's daily values were averaged over each week.
Time Frame: Pre-dose at Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter per minute
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 16 | 17 | 32 | 16
liter per minute
  Morning PEFR: Baseline (n= 16, 17, 32, 16) | 220.0 (113.0) | 236.4 (121.4) | 213.6 (72.6) | 191.0 (77.8)
  Morning PEFR: Change at Week 1 (n= 16, 17, 32, 16) | -3.6 (17.5) | 3.5 (17.8) | 2.1 (13.9) | 1.1 (23.0)
  Morning PEFR: Change at Week 2 (n= 16, 17, 32, 16) | -5.0 (21.0) | -6.0 (18.6) | -1.3 (21.3) | 0.7 (27.2)
  Morning PEFR: Change at Week 3 (n= 15, 17, 31, 16) | -8.8 (27.5) | -6.2 (17.8) | 1.9 (26.4) | 2.6 (22.4)
  Morning PEFR: Change at Week 4 (n= 15, 17, 31, 16) | -5.9 (24.2) | -2.8 (18.4) | 3.3 (31.2) | 2.8 (28.9)
  Morning PEFR: Change at Week 5 (n= 15, 17, 30, 16) | -13.4 (27.2) | -4.4 (21.5) | -9.4 (27.5) | 5.7 (31.0)
  Morning PEFR: Change at Week 6 (n= 15, 17, 30, 15) | -10.5 (27.2) | -4.9 (21.0) | -3.9 (36.6) | -6.1 (26.8)
  Morning PEFR: Change at Week 7 (n= 15, 16, 29, 15) | -8.3 (22.1) | -0.0 (24.3) | 1.2 (33.7) | -2.8 (26.7)
  Morning PEFR: Change at Week 8 (n= 15, 16, 27, 15) | -9.5 (26.8) | -6.8 (29.4) | 0.4 (30.2) | 0.8 (23.1)
  Evening PEFR: Baseline (n= 16, 17, 32, 16) | 242.9 (111.8) | 269.3 (123.1) | 250.0 (78.7) | 207.1 (88.2)
  Evening PEFR: Change at Week 1 (n= 16, 17, 32, 16) | 5.5 (20.5) | -0.2 (16.8) | 3.2 (19.7) | 5.2 (19.5)
  Evening PEFR: Change at Week 2 (n= 16, 17, 32, 16) | 4.8 (27.1) | -8.7 (19.6) | 0.4 (25.9) | 8.5 (37.8)
  Evening PEFR: Change at Week 3 (n= 15, 17, 31, 16) | 0.1 (16.2) | -17.0 (28.6) | 1.6 (22.9) | 7.6 (27.7)
  Evening PEFR: Change at Week 4 (n= 15, 17, 31, 16) | -1.5 (21.5) | -13.7 (19.3) | -0.7 (23.6) | 1.6 (28.5)
  Evening PEFR: Change at Week 5 (n= 15, 17, 30, 16) | -5.4 (23.6) | -14.2 (24.7) | -8.6 (27.0) | 9.5 (36.7)
  Evening PEFR: Change at Week 6 (n= 15, 17, 30, 15) | -5.5 (26.8) | -13.6 (23.2) | -7.3 (27.7) | -4.5 (40.2)
  Evening PEFR: Change at Week 7 (n= 15, 16, 30, 15) | 0.8 (23.7) | -10.7 (21.6) | -6.0 (30.7) | -1.0 (34.5)
  Evening PEFR: Change at Week 8 (n= 15, 16, 28, 15) | -2.6 (21.9) | -16.0 (23.4) | -3.4 (30.6) | -5.9 (41.9)
Statistical Analysis 1: Comparison: UK-432,097 150 Mcg vs Placebo; Morning PEFR, Change at Week 1: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.7292, Mixed Models Analysis; Adjusted Mean Difference = -3.8, 95% CI 1-sided [lower limit -14.3], Standard Error of Mean 6.3
Statistical Analysis 2: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.2768, Mixed Models Analysis; Adjusted Mean Difference = 3.7, 95% CI 1-sided [lower limit -6.6], Standard Error of Mean 6.2
Statistical Analysis 3: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.3795, Mixed Models Analysis; Adjusted Mean Difference = 1.7, 95% CI 1-sided [lower limit -7.4], Standard Error of Mean 5.4
Statistical Analysis 4: Comparison: UK-432,097 150 Mcg vs Placebo; Morning PEFR, Change at Week 2: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.7374, Mixed Models Analysis; Adjusted Mean Difference = -4.9, 95% CI 1-sided [lower limit -17.7], Standard Error of Mean 7.7
Statistical Analysis 5: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 4]; Test type: Superiority or Other; p = 0.7615, Mixed Models Analysis; Adjusted Mean Difference = -5.4, 95% CI 1-sided [lower limit -18.1], Standard Error of Mean 7.6
Statistical Analysis 6: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 4]; Test type: Superiority or Other; p = 0.5811, Mixed Models Analysis; Adjusted Mean Difference = -1.4, 95% CI 1-sided [lower limit -12.4], Standard Error of Mean 6.6
Statistical Analysis 7: Comparison: UK-432,097 150 Mcg vs Placebo; Morning PEFR, Change at Week 3: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.8939, Mixed Models Analysis; Adjusted Mean Difference = -10.9, 95% CI 1-sided [lower limit -25.3], Standard Error of Mean 8.6
Statistical Analysis 8: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p = 0.8117, Mixed Models Analysis; Adjusted Mean Difference = -7.5, 95% CI 1-sided [lower limit -21.6], Standard Error of Mean 8.4
Statistical Analysis 9: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p = 0.4393, Mixed Models Analysis; Adjusted Mean Difference = 1.1, 95% CI 1-sided [lower limit -11.2], Standard Error of Mean 7.4
Statistical Analysis 10: Comparison: UK-432,097 150 Mcg vs Placebo; Morning PEFR, Change at Week 4: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.8055, Mixed Models Analysis; Adjusted Mean Difference = -8.5, 95% CI 1-sided [lower limit -24.7], Standard Error of Mean 9.8
Statistical Analysis 11: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 10]; Test type: Superiority or Other; p = 0.6767, Mixed Models Analysis; Adjusted Mean Difference = -4.4, 95% CI 1-sided [lower limit -20.2], Standard Error of Mean 9.5
Statistical Analysis 12: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 10]; Test type: Superiority or Other; p = 0.4070, Mixed Models Analysis; Adjusted Mean Difference = 2.0, 95% CI 1-sided [lower limit -12.0], Standard Error of Mean 8.4
Statistical Analysis 13: Comparison: UK-432,097 150 Mcg vs Placebo; Morning PEFR, Change at Week 5: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.9705, Mixed Models Analysis; Adjusted Mean Difference = -18.6, 95% CI 1-sided [lower limit -34.7], Standard Error of Mean 9.7
Statistical Analysis 14: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 13]; Test type: Superiority or Other; p = 0.8249, Mixed Models Analysis; Adjusted Mean Difference = -8.9, 95% CI 1-sided [lower limit -24.6], Standard Error of Mean 9.4
Statistical Analysis 15: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 13]; Test type: Superiority or Other; p = 0.9345, Mixed Models Analysis; Adjusted Mean Difference = -12.7, 95% CI 1-sided [lower limit -26.6], Standard Error of Mean 8.3
Statistical Analysis 16: Comparison: UK-432,097 150 Mcg vs Placebo; Morning PEFR, Change at Week 6: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.7384, Mixed Models Analysis; Adjusted Mean Difference = -7.0, 95% CI 1-sided [lower limit -25.3], Standard Error of Mean 11.0
Statistical Analysis 17: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 16]; Test type: Superiority or Other; p = 0.5239, Mixed Models Analysis; Adjusted Mean Difference = -0.6, 95% CI 1-sided [lower limit -18.4], Standard Error of Mean 10.7
Statistical Analysis 18: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 16]; Test type: Superiority or Other; p = 0.4170, Mixed Models Analysis; Adjusted Mean Difference = 2.0, 95% CI 1-sided [lower limit -13.7], Standard Error of Mean 9.4
Statistical Analysis 19: Comparison: UK-432,097 150 Mcg vs Placebo; Morning PEFR, Change at Week 7: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.7695, Mixed Models Analysis; Adjusted Mean Difference = -7.6, 95% CI 1-sided [lower limit -24.8], Standard Error of Mean 10.3
Statistical Analysis 20: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 19]; Test type: Superiority or Other; p = 0.4566, Mixed Models Analysis; Adjusted Mean Difference = 1.1, 95% CI 1-sided [lower limit -15.6], Standard Error of Mean 10.1
Statistical Analysis 21: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 19]; Test type: Superiority or Other; p = 0.3535, Mixed Models Analysis; Adjusted Mean Difference = 3.3, 95% CI 1-sided [lower limit -11.4], Standard Error of Mean 8.9
Statistical Analysis 22: Comparison: UK-432,097 150 Mcg vs Placebo; Morning PEFR, Change at Week 8: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.8598, Mixed Models Analysis; Adjusted Mean Difference = -12.1, 95% CI 1-sided [lower limit -30.7], Standard Error of Mean 11.1
Statistical Analysis 23: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 22]; Test type: Superiority or Other; p = 0.8005, Mixed Models Analysis; Adjusted Mean Difference = -9.2, 95% CI 1-sided [lower limit -27.4], Standard Error of Mean 10.9
Statistical Analysis 24: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 22]; Test type: Superiority or Other; p = 0.3441, Mixed Models Analysis; Adjusted Mean Difference = 3.9, 95% CI 1-sided [lower limit -12.2], Standard Error of Mean 9.6
Statistical Analysis 25: Comparison: UK-432,097 150 Mcg vs Placebo; Evening PEFR, Change at Week 1: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.4436, Mixed Models Analysis; Adjusted Mean Difference = 1.0, 95% CI 1-sided [lower limit -10.5], Standard Error of Mean 6.9
Statistical Analysis 26: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 25]; Test type: Superiority or Other; p = 0.7238, Mixed Models Analysis; Adjusted Mean Difference = -4.1, 95% CI 1-sided [lower limit -15.5], Standard Error of Mean 6.8
Statistical Analysis 27: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 25]; Test type: Superiority or Other; p = 0.5743, Mixed Models Analysis; Adjusted Mean Difference = -1.1, 95% CI 1-sided [lower limit -11.1], Standard Error of Mean 6.0
Statistical Analysis 28: Comparison: UK-432,097 150 Mcg vs Placebo; Evening PEFR, Change at Week 2: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.6190, Mixed Models Analysis; Adjusted Mean Difference = -3.0, 95% CI 1-sided [lower limit -19.3], Standard Error of Mean 9.8
Statistical Analysis 29: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 28]; Test type: Superiority or Other; p = 0.9473, Mixed Models Analysis; Adjusted Mean Difference = -15.9, 95% CI 1-sided [lower limit -32.1], Standard Error of Mean 9.7
Statistical Analysis 30: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 28]; Test type: Superiority or Other; p = 0.8014, Mixed Models Analysis; Adjusted Mean Difference = -7.3, 95% CI 1-sided [lower limit -21.4], Standard Error of Mean 8.5
Statistical Analysis 31: Comparison: UK-432,097 150 Mcg vs Placebo; Evening PEFR, Change at Week 3: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.7929, Mixed Models Analysis; Adjusted Mean Difference = -7.1, 95% CI 1-sided [lower limit -21.5], Standard Error of Mean 8.6
Statistical Analysis 32: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 31]; Test type: Superiority or Other; p = 0.9963, Mixed Models Analysis; Adjusted Mean Difference = -23.2, 95% CI 1-sided [lower limit -37.3], Standard Error of Mean 8.4
Statistical Analysis 33: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 31]; Test type: Superiority or Other; p = 0.7387, Mixed Models Analysis; Adjusted Mean Difference = -4.8, 95% CI 1-sided [lower limit -17.1], Standard Error of Mean 7.4
Statistical Analysis 34: Comparison: UK-432,097 150 Mcg vs Placebo; Evening PEFR, Change at Week 4: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.6286, Mixed Models Analysis; Adjusted Mean Difference = -2.8, 95% CI 1-sided [lower limit -16.8], Standard Error of Mean 8.4
Statistical Analysis 35: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 34]; Test type: Superiority or Other; p = 0.9538, Mixed Models Analysis; Adjusted Mean Difference = -14.1, 95% CI 1-sided [lower limit -27.8], Standard Error of Mean 8.3
Statistical Analysis 36: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 34]; Test type: Superiority or Other; p = 0.5701, Mixed Models Analysis; Adjusted Mean Difference = -1.3, 95% CI 1-sided [lower limit -13.4], Standard Error of Mean 7.3
Statistical Analysis 37: Comparison: UK-432,097 150 Mcg vs Placebo; Evening PEFR, Change at Week 5: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.9242, Mixed Models Analysis; Adjusted Mean Difference = -14.5, 95% CI 1-sided [lower limit -31.3], Standard Error of Mean 10.0
Statistical Analysis 38: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 37]; Test type: Superiority or Other; p = 0.9876, Mixed Models Analysis; Adjusted Mean Difference = -22.4, 95% CI 1-sided [lower limit -38.8], Standard Error of Mean 9.8
Statistical Analysis 39: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 37]; Test type: Superiority or Other; p = 0.9802, Mixed Models Analysis; Adjusted Mean Difference = -18.1, 95% CI 1-sided [lower limit -32.5], Standard Error of Mean 8.7
Statistical Analysis 40: Comparison: UK-432,097 150 Mcg vs Placebo; Evening PEFR, Change at Week 6: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.5705, Mixed Models Analysis; Adjusted Mean Difference = -1.9, 95% CI 1-sided [lower limit -19.5], Standard Error of Mean 10.6
Statistical Analysis 41: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 40]; Test type: Superiority or Other; p = 0.8063, Mixed Models Analysis; Adjusted Mean Difference = -9.0, 95% CI 1-sided [lower limit -26.1], Standard Error of Mean 10.3
Statistical Analysis 42: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 40]; Test type: Superiority or Other; p = 0.6667, Mixed Models Analysis; Adjusted Mean Difference = -3.9, 95% CI 1-sided [lower limit -19.1], Standard Error of Mean 9.1
Statistical Analysis 43: Comparison: UK-432,097 150 Mcg vs Placebo; Evening PEFR, Change at Week 7: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.4640, Mixed Models Analysis; Adjusted Mean Difference = 0.9, 95% CI 1-sided [lower limit -16.4], Standard Error of Mean 10.4
Statistical Analysis 44: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 43]; Test type: Superiority or Other; p = 0.8821, Mixed Models Analysis; Adjusted Mean Difference = -12.2, 95% CI 1-sided [lower limit -29.3], Standard Error of Mean 10.2
Statistical Analysis 45: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 43]; Test type: Superiority or Other; p = 0.7591, Mixed Models Analysis; Adjusted Mean Difference = -6.4, 95% CI 1-sided [lower limit -21.4], Standard Error of Mean 9.0
Statistical Analysis 46: Comparison: UK-432,097 150 Mcg vs Placebo; Evening PEFR, Change at Week 8: Analysis was performed using longitudinal mixed effect model with baseline value, treatment, week, and treatment by week as fixed effects and participants as random effect; Test type: Superiority or Other; p = 0.4001, Mixed Models Analysis; Adjusted Mean Difference = 2.8, 95% CI 1-sided [lower limit -15.6], Standard Error of Mean 11.0
Statistical Analysis 47: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 17, analysis 46]; Test type: Superiority or Other; p = 0.8707, Mixed Models Analysis; Adjusted Mean Difference = -12.3, 95% CI 1-sided [lower limit -30.3], Standard Error of Mean 10.8
Statistical Analysis 48: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 17, analysis 46]; Test type: Superiority or Other; p = 0.4629, Mixed Models Analysis; Adjusted Mean Difference = 0.9, 95% CI 1-sided [lower limit -15.0], Standard Error of Mean 9.6

18. Secondary Outcome: Number of Participants With Categorical Scores on Clinical Global Impression of Change (CGI-C)
Description: CGI-C: clinician's global impression of a participant's clinical condition in terms of change relative to the start of treatment. Rated on a 7-point scale from 1 (very much improved) to 7 (very much worse). Higher score = more affected.
Time Frame: Week 6
Population: FAS: all randomized participants, who received at least 2 weeks of dosing and had at least 1 valid FEV1 measurement during treatment. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 14 | 16 | 29 | 15
participants
  Very Much Improved | 0 | 0 | 0 | 1
  Much Improved | 0 | 2 | 2 | 2
  Minimally Improved | 5 | 4 | 9 | 4
  No Change | 5 | 7 | 14 | 6
  Minimally Worse | 2 | 3 | 4 | 2
  Much Worse | 2 | 0 | 0 | 0
  Very Much Worse | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: UK-432,097 150 Mcg vs Placebo; A proportional odds model was fitted using Proc Logistic in Statistical Analysis System (SAS), using treatment as a categorical variable and center as a covariate. The odds ratio and corresponding 95% confidence interval were tested using Type III (Wald) tests; Test type: Superiority or Other; Odds Ratio (OR) = 0.6428, 95% CI 2-sided [0.2023 to 2.0419]
Statistical Analysis 2: Comparison: UK-432,097 450 Mcg vs Placebo; A proportional odds model was fitted using Proc Logistic in SAS, using treatment as a categorical variable and center as a covariate. The odds ratio and corresponding 95% confidence interval were tested using Type III (Wald) tests; Test type: Superiority or Other; Odds Ratio (OR) = 0.5574, 95% CI 2-sided [0.1505 to 2.0647]
Statistical Analysis 3: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 18, analysis 2]; Test type: Superiority or Other; Odds Ratio (OR) = 0.3270, 95% CI 2-sided [0.0830 to 1.2879]

19. Secondary Outcome: Number of Participants With Categorical Scores on Patient Global Impression of Change (PGI-C)
Description: PGI-C: participant rated instrument to measure participant's clinical condition in terms of change relative to the start of treatment. Rated on a 7-point scale from 1 (very much improved) to 7 (very much worse). Higher score = more affected.
Time Frame: Week 6
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 14 | 16 | 29 | 15
participants
  Very Much Improved | 0 | 0 | 0 | 0
  Much Improved | 2 | 2 | 3 | 2
  Minimally Improved | 3 | 4 | 7 | 6
  No Change | 7 | 8 | 15 | 5
  Minimally Worse | 1 | 1 | 2 | 2
  Much Worse | 1 | 0 | 1 | 0
  Very Much Worse | 0 | 1 | 1 | 0
Statistical Analysis 1: Comparison: UK-432,097 150 Mcg vs Placebo; [analysis description as in outcome 18, analysis 2]; Test type: Superiority or Other; Odds Ratio (OR) = 0.5709, 95% CI 2-sided [0.1790 to 1.8204]
Statistical Analysis 2: Comparison: UK-432,097 450 Mcg vs Placebo; [analysis description as in outcome 18, analysis 2]; Test type: Superiority or Other; Odds Ratio (OR) = 0.6416, 95% CI 2-sided [0.1736 to 2.3715]
Statistical Analysis 3: Comparison: UK-432,097 1350 Mcg vs Placebo; [analysis description as in outcome 18, analysis 2]; Test type: Superiority or Other; Odds Ratio (OR) = 0.5877, 95% CI 2-sided [0.1516 to 2.2777]

20. Other Pre Specified Outcome: Change From Baseline in Pulse Rate at Week 0, 1, 2, 4, and 6
Description: Pulse rate: the number of pulsations noted in a peripheral artery per unit of time after participant rested supine for 5 minutes, reported as beats per minute (bpm).
Time Frame: Baseline (pre-dose at Week 0); Pre-dose and 3-hour post-dose on Week 1, 6; 3-hour post-dose on Week 0, 2, 4
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. Here "n" signifies participants who were evaluable for specified time-point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 17 | 18 | 35 | 17
bpm
  Baseline (n= 17, 18, 35, 17) | 68.6 (11.45) | 75.2 (12.37) | 73.7 (12.83) | 74.2 (13.07)
  Change at Week 0, Post-Dose (n= 16, 18, 35, 17) | -0.4 (6.86) | 2.5 (6.72) | 1.3 (7.63) | 0.3 (7.86)
  Change at Week 1, Pre-Dose (n= 15, 18, 33, 16) | 3.2 (7.97) | 4.7 (10.97) | 0.8 (9.95) | -0.3 (10.10)
  Change at Week 1, Post-Dose (n= 17, 15, 32, 16) | 2.7 (10.10) | 2.2 (7.47) | 1.1 (8.91) | 0.5 (10.47)
  Change at Week 2, Post-Dose (n= 16, 17, 30, 16) | 1.6 (9.04) | -1.7 (10.80) | 2.7 (12.39) | 0.1 (6.97)
  Change at Week 4, Post-Dose (n= 15, 15, 30, 16) | 2.5 (10.08) | 1.3 (10.15) | 3.8 (16.52) | 2.4 (7.73)
  Change at Week 6, Pre-Dose (n= 15, 16, 28, 15) | 0.7 (6.16) | -0.1 (6.70) | 0.9 (11.39) | -1.2 (6.57)
  Change at Week 6, Post-Dose (n= 14, 16, 28, 15) | 2.2 (8.23) | -0.2 (7.44) | 3.5 (12.85) | 1.2 (8.88)

21. Other Pre Specified Outcome: Change From Baseline in Blood Pressure at Week 0, 1, 2, 4, and 6
Description: BP is the pressure of the blood within the arteries. It is produced primarily by the contraction of the heart muscle. BP measurement is recorded by 2 numbers: systolic BP (SBP, BP when heart is contracting; it is the maximum arterial pressure during contraction of left ventricle) and diastolic BP (DBP, BP when heart is relaxing; it is the minimum arterial pressure during relaxation and dilation of ventricles). BP was measured by sphygmomanometer (manual or semi-automated) using appropriate-sized and calibrated cuff after participant rested in supine position for 5 minutes.
Time Frame: Baseline (pre-dose at Week 0); Pre-dose and 3-hour post-dose on Week 1, 6; 3-hour post-dose on Week 0, 2, 4
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 17 | 18 | 35 | 17
millimeter of mercury (mmHg)
  SBP: Baseline (n= 17, 18, 35, 17) | 128.5 (11.73) | 137.3 (14.40) | 129.5 (12.77) | 132.7 (13.45)
  SBP: Change at Week 0, Post-Dose (n= 16,18,35,17) | 2.4 (7.29) | -1.3 (11.52) | -1.3 (9.70) | 0.4 (7.36)
  SBP: Change at Week 1, Pre-Dose (n= 15,18,33,16) | 1.4 (6.33) | -1.4 (15.34) | 0.7 (12.32) | 0.3 (11.98)
  SBP: Change at Week 1, Post-Dose (n= 17,15,32,16) | 0.5 (9.90) | -5.5 (16.17) | 1.0 (15.41) | -4.5 (12.81)
  SBP: Change at Week 2, Post-Dose (n= 16,17,30,16) | 1.4 (16.25) | 2.8 (16.64) | 0.5 (13.06) | -2.2 (14.86)
  SBP: Change at Week 4, Post-Dose (n= 15,15,30,16) | 3.1 (6.27) | -4.7 (12.96) | -1.3 (14.56) | -5.8 (15.21)
  SBP: Change at Week 6, Pre-Dose (n= 15,16,28,15) | 3.6 (11.57) | -7.6 (15.19) | -1.5 (9.54) | 1.2 (10.81)
  SBP: Change at Week 6, Post-Dose (n= 14,16,28,15) | -1.2 (10.14) | -7.5 (13.73) | -0.9 (8.77) | -0.9 (12.68)
  DBP: Baseline (n= 17, 18, 35, 17) | 76.9 (7.18) | 78.5 (10.29) | 74.3 (8.30) | 76.5 (7.24)
  DBP: Change at Week 0, Post-Dose (n= 16,18,35,17) | 0.1 (5.97) | -2.0 (6.21) | -0.7 (6.30) | 0.6 (6.44)
  DBP: Change at Week 1, Pre-Dose (n= 15,18,33,16) | 1.1 (10.56) | -0.8 (6.18) | -0.1 (8.68) | 1.5 (6.23)
  DBP: Change at Week 1, Post-Dose (n= 17,15,32,16) | -1.9 (9.86) | -2.1 (8.72) | -0.2 (8.95) | -1.0 (7.41)
  DBP: Change at Week 2, Post-Dose (n= 16,17,30,16) | -0.6 (11.28) | 0.1 (7.96) | -0.5 (8.07) | 0.1 (7.64)
  DBP: Change at Week 4, Post-Dose (n= 15,15,30,16) | -1.8 (7.53) | -4.5 (6.49) | -1.9 (8.10) | -1.2 (7.79)
  DBP: Change at Week 6, Pre-Dose (n= 15,16,28,15) | -2.2 (6.28) | -3.9 (8.21) | -0.3 (6.74) | 0.7 (5.09)
  DBP: Change at Week 6, Post-Dose (n= 14,16,28,15) | -5.2 (6.90) | -7.3 (7.88) | -2.8 (6.87) | -3.5 (8.27)

22. Other Pre Specified Outcome: Change From Baseline in 12-Lead Electrocardiogram (ECG) Parameters (QT, QTc, QTcB, QTcF, QRS, RR and PR) at Week 0, 1, 2, 4, 6, and 8
Description: Standard 12-lead ECG was performed after participant has rested for at least 10 minutes in supine position. ECG intervals (Int) included PR Int (time between onset of atrial depolarization and onset of ventricular depolarization), QRS Int (represented ventricular depolarization), RR Int (time between 2 QRS complex), QT Int (time corresponding to the beginning of depolarization to repolarization of the ventricles), corrected QT (QTc) Int, QT Int corrected by Fridericia's formula (QTcF=QT divided by cube root of RR Int) and Bazett's formula (QTcB=QT divided by square root of RR Int).
Time Frame: Baseline (pre-dose at Week 0); Pre-dose and 3-hour post-dose on Week 6; 3-hour post-dose on Week 0, 1, 2, 4; Week 8 (follow-up)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 17 | 18 | 35 | 17
milliseconds (msec)
  RR: Baseline (n= 17,18,34,17) | 747.0 (351.66) | 696.1 (357.91) | 733.3 (281.12) | 745.7 (362.90)
  RR: Change at Week 0, Post-Dose (n= 17,18,34,17) | 34.4 (174.39) | -63.7 (82.96) | -2.0 (100.92) | -6.1 (93.51)
  RR: Change at Week 1, Post-Dose (n= 17,17,31,16) | 45.8 (250.92) | -62.8 (82.17) | 7.3 (112.16) | 6.0 (113.17)
  RR: Change at Week 2, Post-Dose (n= 16,17,31,16) | -18.5 (111.03) | -49.1 (131.10) | 12.0 (120.00) | -78.6 (202.34)
  RR: Change at Week 4, Post-Dose (n= 15,17,28,16) | 98.1 (291.65) | -88.7 (194.50) | -6.6 (144.20) | -66.0 (196.32)
  RR: Change at Week 6, Pre-Dose (n= 14,16,28,15) | -19.3 (72.80) | -32.3 (84.20) | -1.6 (101.00) | -24.6 (206.21)
  RR: Change at Week 6, Post-Dose (n= 15,16,27,15) | -22.9 (109.20) | -43.7 (99.03) | -27.3 (124.20) | -34.9 (233.38)
  RR: Change at Week 8 (n= 17,18,31,17) | -10.4 (85.52) | -36.4 (83.34) | -1.1 (185.33) | -19.3 (200.12)
  PR: Baseline (n= 17,18,35,17) | 165.6 (23.91) | 165.0 (23.03) | 171.2 (26.92) | 172.8 (23.89)
  PR: Change at Week 0, Post-Dose (n= 17,18,35,17) | -0.7 (6.85) | -1.3 (8.51) | -2.4 (8.59) | 0.8 (16.21)
  PR: Change at Week 1, Post-Dose (n= 17,17,32,16) | 2.0 (12.43) | -0.6 (13.79) | 2.0 (19.93) | 0.2 (22.78)
  PR: Change at Week 2, Post-Dose (n= 16,17,32,16) | 1.6 (14.30) | 1.1 (13.33) | -4.1 (11.34) | 6.4 (40.37)
  PR: Change at Week 4, Post-Dose (n= 15,17,29,16) | 2.8 (11.81) | -2.5 (11.93) | 6.5 (49.74) | 9.2 (37.48)
  PR: Change at Week 6, Pre-Dose (n= 14,16,29,15) | -2.4 (10.11) | 2.4 (12.85) | -2.1 (10.59) | 0.2 (26.08)
  PR: Change at Week 6, Post-Dose (n= 15,16,28,15) | -1.5 (14.85) | 1.9 (14.63) | -3.0 (13.56) | 4.4 (29.21)
  PR: Change at Week 8 (n= 17,18,32,17) | -4.9 (16.05) | -2.2 (13.17) | -3.6 (13.71) | -0.4 (16.64)
  QRS: Baseline (n= 17,18,35,17) | 93.2 (10.58) | 89.1 (11.40) | 85.8 (26.19) | 92.7 (14.93)
  QRS: Change at Week 0, Post-Dose (n= 17,18,35,17) | -0.4 (4.49) | 0.9 (3.31) | -1.0 (5.52) | -2.1 (9.82)
  QRS: Change at Week 1, Post-Dose (n= 17,17,32,16) | -1.7 (12.30) | -0.6 (5.70) | -1.7 (6.11) | 5.6 (28.56)
  QRS: Change at Week 2, Post-Dose (n= 16,17,32,16) | -0.2 (6.92) | 2.3 (4.96) | -2.6 (8.15) | -4.6 (9.82)
  QRS: Change at Week 4, Post-Dose (n= 15,17,29,16) | -0.2 (5.95) | -0.7 (9.40) | -0.9 (6.30) | -2.2 (12.45)
  QRS: Change at Week 6, Pre-Dose (n= 14,16,29,15) | 2.2 (5.30) | -1.4 (7.54) | -2.5 (7.37) | -4.2 (10.91)
  QRS: Change at Week 6, Post-Dose (n= 15,16,28,15) | 3.4 (6.00) | -1.4 (9.70) | -1.3 (5.94) | -4.3 (10.86)
  QRS: Change at Week 8 (n= 17,18,32,17) | 0.5 (5.58) | 0.8 (3.88) | 0.1 (8.09) | -4.0 (9.02)
  QT: Baseline (n= 17,18,35,17) | 387.9 (27.09) | 384.0 (37.04) | 371.9 (27.52) | 381.7 (40.08)
  QT: Change at Week 0, Post-Dose (n= 17,18,35,17) | 3.2 (16.81) | -5.1 (10.90) | 5.6 (22.76) | 1.4 (22.92)
  QT: Change at Week 1, Post-Dose (n= 17,17,32,16) | -1.8 (27.75) | -12.5 (16.61) | 6.4 (23.75) | 1.6 (29.10)
  QT: Change at Week 2, Post-Dose (n= 16,17,32,16) | 15.4 (66.03) | -5.1 (18.91) | 3.4 (28.34) | 2.0 (26.65)
  QT: Change at Week 4, Post-Dose (n= 15,17,29,16) | 0.2 (25.61) | -3.9 (19.91) | 6.5 (36.69) | -1.6 (29.41)
  QT: Change at Week 6, Pre-Dose (n= 14,16,29,15) | 6.6 (21.85) | -5.0 (16.06) | 6.3 (25.40) | 2.6 (22.65)
  QT: Change at Week 6, Post-Dose (n= 15,16,28,15) | 9.7 (30.00) | -3.6 (17.51) | 5.0 (30.17) | 3.4 (28.95)
  QT: Change at Week 8 (n= 17,18,32,17) | 5.3 (26.56) | -6.8 (20.08) | 11.3 (23.65) | -0.5 (18.66)
  QTc: Baseline (n= 17,18,35,17) | 401.1 (22.91) | 409.6 (20.70) | 409.2 (25.92) | 410.8 (20.63)
  QTc: Change at Week 0, Post-Dose (n= 17,18,35,17) | 6.9 (11.00) | 7.1 (14.01) | 7.1 (20.17) | 4.3 (14.15)
  QTc: Change at Week 1, Post-Dose (n= 17,17,32,16) | -2.1 (22.79) | -0.0 (10.52) | 3.3 (23.46) | 3.5 (10.63)
  QTc: Change at Week 2, Post-Dose (n= 16,17,32,16) | 18.5 (58.27) | 4.8 (19.04) | 3.0 (21.77) | 5.8 (22.96)
  QTc: Change at Week 4, Post-Dose (n= 15,17,29,16) | 1.6 (20.58) | 5.5 (18.94) | 9.4 (26.13) | 3.8 (23.36)
  QTc: Change at Week 6, Pre-Dose (n= 14,16,29,15) | 12.4 (16.86) | -0.4 (9.68) | 8.5 (22.91) | -4.7 (16.79)
  QTc: Change at Week 6, Post-Dose (n= 15,16,28,15) | 15.0 (15.87) | 5.4 (16.94) | 10.6 (24.11) | -1.6 (20.10)
  QTc: Change at Week 8 (n= 17,18,32,17) | 11.5 (23.83) | 0.1 (10.34) | 9.1 (25.30) | -8.8 (15.00)
  QTcB: Baseline (n= 17,18,35,17) | 405.7 (27.46) | 417.2 (18.69) | 412.0 (25.85) | 413.6 (18.26)
  QTcB: Change at Week 0, Post-Dose (n= 17,18,35,17) | 6.7 (11.69) | 6.8 (12.56) | 7.2 (21.29) | 9.8 (14.48)
  QTcB: Change at Week 1, Post-Dose (n= 17,17,32,16) | 0.9 (16.06) | -0.3 (14.53) | 4.2 (24.27) | 7.8 (17.50)
  QTcB: Change at Week 2, Post-Dose (n= 16,17,32,16) | 17.9 (56.34) | 7.6 (16.39) | 4.1 (23.21) | 8.5 (18.05)
  QTcB: Change at Week 4, Post-Dose (n= 15,17,29,16) | -0.7 (24.27) | 4.0 (13.95) | 11.3 (29.54) | 9.2 (18.59)
  QTcB: Change at Week 6, Pre-Dose (n= 14,16,29,15) | 13.0 (14.92) | -1.0 (12.81) | 10.0 (24.00) | -1.5 (12.18)
  QTcB: Change at Week 6, Post-Dose (n= 15,16,28,15) | 15.2 (13.76) | 3.8 (16.69) | 13.9 (23.88) | 3.0 (11.68)
  QTcB: Change at Week 8 (n= 17,18,32,17) | 11.6 (24.91) | -1.2 (10.21) | 10.7 (28.23) | -6.2 (13.54)
  QTcF: Baseline (n= 17,18,35,17) | 399.4 (22.33) | 405.4 (22.06) | 397.8 (20.90) | 402.3 (20.33)
  QTcF: Change at Week 0, Post-Dose (n= 17,18,35,17) | 5.5 (10.29) | 2.8 (9.30) | 6.7 (19.10) | 6.8 (15.06)
  QTcF: Change at Week 1, Post-Dose (n= 17,17,32,16) | -0.1 (16.61) | -4.5 (12.73) | 5.2 (20.60) | 5.4 (15.26)
  QTcF: Change at Week 2, Post-Dose (n= 16,17,32,16) | 16.9 (58.63) | 3.1 (11.21) | 4.1 (20.59) | 6.2 (18.85)
  QTcF: Change at Week 4, Post-Dose (n= 15,17,29,16) | -0.4 (21.21) | 1.3 (12.14) | 9.4 (27.88) | 5.6 (20.76)
  QTcF: Change at Week 6, Pre-Dose (n= 14,16,29,15) | 10.9 (16.11) | -2.4 (9.75) | 8.8 (20.37) | -0.0 (13.67)
  QTcF: Change at Week 6, Post-Dose (n= 15,16,28,15) | 13.2 (17.11) | 1.3 (14.15) | 10.9 (22.53) | 3.1 (14.58)
  QTcF: Change at Week 8 (n= 17,18,32,17) | 9.4 (24.35) | -3.0 (10.38) | 10.9 (23.31) | -4.3 (10.00)

23. Other Pre Specified Outcome: Change From Baseline in 12-Lead Electrocardiogram (ECG) Parameters (Heart Rate) at Week 0, 1, 2, 4, 6, and 8
Description: Standard 12-lead ECG was performed after the participant has rested quietly for at least 10 minutes in supine position. The time interval between consecutive heart beats (RR interval) was used to calculate heart rate.
Time Frame: as for outcome 22
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 17 | 18 | 35 | 17
bpm
  Baseline (n= 17,18,35,17) | 66.6 (11.65) | 72.1 (11.00) | 74.8 (12.92) | 72.4 (13.81)
  Change at Week 0, Post-Dose (n= 17,18,35,17) | 0.8 (6.56) | 4.0 (5.90) | 0.3 (8.69) | 2.7 (7.76)
  Change at Week 1, Post-Dose (n= 17,17,32,16) | 1.1 (9.76) | 4.3 (6.30) | -1.5 (10.13) | 2.8 (13.45)
  Change at Week 2, Post-Dose (n= 16,17,32,16) | 0.7 (8.98) | 4.2 (10.38) | -0.2 (12.76) | 1.9 (8.06)
  Change at Week 4, Post-Dose (n= 15,17,29,16) | -0.2 (8.75) | 2.4 (8.33) | 2.5 (18.51) | 3.2 (8.23)
  Change at Week 6, Pre-Dose (n= 14,16,29,15) | 2.3 (5.17) | 1.4 (7.71) | 0.6 (11.82) | -1.7 (7.72)
  Change at Week 6, Post-Dose (n= 15,16,28,15) | 1.9 (8.68) | 2.2 (6.94) | 2.6 (11.84) | 0.3 (11.31)
  Change at Week 8 (n= 17,18,32,17) | 1.9 (5.94) | 1.8 (6.51) | -0.8 (11.16) | -2.1 (9.57)

24. Other Pre Specified Outcome: Change in Post-Study Drug Forced Expiratory Volume in 1 Second (FEV1) Compared to Pre-Study Drug Forced Expiratory Volume in 1 Second (FEV1) at Week 0, 1, 2, 4, and 6
Description: FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Post-study drug FEV1 was obtained from spirometry, performed 15-30 minutes after study treatment administration. Pre-study drug FEV1 was obtained from spirometry, performed before study treatment administration.
Time Frame: Pre-dose and 15 to 30 minutes Post-dose at Week 0, 1, 2, 4, 6
Population: Data for this pre-specified endpoint was not analyzed, as the study was terminated due to futility based on results of interim analysis.
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | UK-432,097 150 Mcg | UK-432,097 450 Mcg | UK-432,097 1350 Mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18 | 0/35 | 0/17
Other Adverse Events (participants affected / at risk) | 11/17 | 8/18 | 11/35 | 10/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UK-432,097 150 Mcg (N=17) | UK-432,097 450 Mcg (N=18) | UK-432,097 1350 Mcg (N=35) | Placebo (N=17)
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 2 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 2 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 3 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0
Forced expiratory volume decreased (Investigations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Study was terminated prematurely due to futility based on results of interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.